CLINICAL TRIAL: NCT04778826
Title: Immune Response of Patients Following Thoracoscopic Lobectomy Along With Bilateral Transcervical Mediastinal Lymphadenectomy and Patients Receiving VATSLOB Together With Standard Unilateral Mediastinal Lymphadenectomy
Brief Title: Immune Response Following Lobectomy Along With or Without Bilateral Transcervical Mediastinal Lymphadenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Otto Wagner Hospital (Other)
Collaborators: Medtronic Spine LLC (Industry)
Responsible Party: Principal Investigator, Mohamed Salama, Clinical Professor, Otto Wagner Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: combined Lobectomy and VAMLA
Record Dates: First submitted 2020-10-15; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Lung Neoplasm Malignant
Keywords: lung lobectomy; lymphadenectomy
MeSH Terms: conditions — Lung Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Intervention Model Description: Compare the oncological outcome and immune competence between patients who undergo lung lobectomy with standard lymphadenectomy and those who undergo combined lobectomy and video assisted bilateral mediastinal lymphadenectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Lobectomy with standard ipsilateral lymphadenectomy (Active Comparator): Lung lobectomy with ipsilateral lymphadenectomy
  Interventions: Procedure: Lymphadenectomy
- Lung Lobectomy with VAMLA (Active Comparator): Lung lobectomy combined with video-assisted mediastinal lymphadenectomy through the neck (VAMLA). The approach is similar to transcervical mediastinoscopy and allows for a radical bloc dissection of all mediastinal lymph node stations. Besides the benefit of bilateral lung ventilation during this phase of the operation a bilateral mediastinal lymphadenectomy offers improved surgical radicality.
  Interventions: Procedure: Lymphadenectomy

INTERVENTIONS:
Procedure: Lymphadenectomy — radical bloc dissection of all mediastinal lymph node stations

SUMMARY:
Any kind of anatomical lung resection for lung cancer with curative intent has to be accompanied by formal mediastinal lymph node dissection. Video-assisted mediastinoscopic lymphadenectomy through a cervical access (VAMLA) along with thoracoscopic lobectomies in the same setting offers improved radicality through bilateral mediastinal dissection, provide accurate staging, does not require single lung ventilation and hence ideally supports the concept of minimally invasive surgery.

Due to the VAMLA associated radicality, the investigator believes that using of VAMLA along with lobectomy could improve the oncological outcome of lung cancer patients. Furthermore, the absence of single lung ventilation during VAMLA could attenuate the surgically induced immunosuppression.

DETAILED DESCRIPTION:
Any kind of anatomical lung resection for lung cancer with curative intent has to be accompanied by formal mediastinal lymph node dissection. Video-assisted mediastinoscopic lymphadenectomy through a cervical access (VAMLA) along with thoracoscopic lobectomies in the same setting offers improved radicality through bilateral mediastinal dissection, provide accurate staging, does not require single lung ventilation and hence ideally supports the concept of minimally invasive surgery.

Due to the VAMLA associated radicality, the investigator believes that using VAMLA along with lobectomy could improve the oncological outcome of lung cancer patients. Furthermore, the absence of single lung ventilation during VAMLA could attenuate the surgically induced immunosuppression.

The present study aims at:

1. The current project primarily aims at identifying the effect of reduced single lunge ventilation time during VAMLA-VATS lobectomy on the intraoperative production of oxygen radicals as well as its effect on the immune competence of patients undergoing VAMLA-VATS lobectomy as compared to those receiving VATS lobectomy Along with conventional unilateral lymphadenectomy.
2. Secondary, in line with the hypothesis that radical bilateral lymphadenectomy might results in a more complete oncological staging as compared to unilateral lymphadenectomy or lymph node sampling. The current project aims to compare the pre- and postoperative staging in patients undergoing VAMLA, as VAMLA enables a proper examination of all bilateral mediastinal lymph nodes.
3. Patient Follow-up will be continued for at least 5 years postoperatively in order to compare the oncological outcome namely local and distant recurrence, tumor-associated and overall survival in patients undergoing VAMLA-VATS Lobectomy as compared to those with VATS lobectomy. This issue is, however, a second endpoint of this study and will be independent of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* adult
* non small cell lung cancer
* operable tumor
* indicated for endoscopic lung surgery

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative interleukins | 1st postoperative day
  Interleukin (IL) 6 serum concentration on the 1st postoperative day

SECONDARY OUTCOMES:
Hospitalisation | until discharge from hospital, assessed up to 14 days
  Discharge from hospital
Overall Survival | 5 years
  5 years survival

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Mueller, MD, Study Director — Department of thoracic Surgery, Clinic Floridsdorf
Locations (1):
- Department of Thoracic Surgery, clinic Floridsdorf, Vienna, Austria

REFERENCES:
- [Derived] Salama M, Mueller MR. Enhanced recovery in lung surgery: coaxial versus conventional chest drains following video-assisted thoracoscopic surgery lobectomy-a prospective randomized trial. J Thorac Dis. 2025 Nov 30;17(11):10262-10271. doi: 10.21037/jtd-2025-1169. Epub 2025 Nov 26. PMID 41376917